CLINICAL TRIAL: NCT06288919
Title: Erythritol vs Ultrasonic Scaler Prophylaxis Systems on Dental Implants With Different Types of Crowns: 24-months Randomized Clinical Trial
Brief Title: Erythritol vs Ultrasonic Scaler Prophylaxis Systems on Dental Implants With Crowns Made by Different Materials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-IMPLHYGIENE
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Dental Implant Failed; Peri-implant Mucositis; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythritol group (Experimental)
  Interventions: Other: Erythritol prophylactic powders
- Ultrasonic scaler (Active Comparator)
  Interventions: Other: Ultrasonic scaler with peek inserts

INTERVENTIONS:
Other: Erythritol prophylactic powders — erythritol with particle size of ~14 µm will be used for 5 seconds (AIRFLOW® PLUS EMS)
  Arms: Erythritol group
Other: Ultrasonic scaler with peek inserts — ultrasonic scaler, a piezoelectric handpiece with peek inserts (Mini Piezon EMS; PI, EMS) will be used.
  Arms: Ultrasonic scaler

SUMMARY:
The aim of the study is to assess which prophylaxis methods is the most suitable for peri-implant hygiene between erythritol and ultrasonic scaler with peek inserts.

A randomized clinical trial will be conducted on the patient. Patients will be randomly divided into two groups:

* Erythritol group: erythritol with a particle size of ~14 µm will be used for 5 seconds (AIRFLOW® PLUS EMS)
* Ultrasonic scaler group: a piezoelectric handpiece with peek inserts (Mini Piezon EMS; PI EMS) will be used.

Different subgroups will be defined according to the material of the dental crown of the related implant.

The oral hygiene session will be carried out every 6 months (2-years follow-up; 6 sessions), after instruction and motivation of the patient, completion of the clinical chart with the recording of the Probing Depth (evaluation in mm of the peri-implant sulcus taken by a periodontal probe; 4 surfaces of the gingival margin are detected: vestibular, palatal/lingual, mesial, distal), Bleeding on Probing and Plaque Index.

DETAILED DESCRIPTION:
The aim of the study is to assess which prophylaxis methods is the most suitable for peri-implant hygiene between erythritol and ultrasonic scaler with peek inserts.

A randomized clinical trial will be conducted on the patient. Patients will be randomly divided into two groups:

* Erythritol group: erythritol with a particle size of ~14 µm will be used for 5 seconds (AIRFLOW® PLUS EMS)
* Ultrasonic scaler group: a piezoelectric handpiece with peek inserts (Mini Piezon EMS; PI EMS) will be used.

Different subgroups will be defined according to the material of the dental crown of the related implant: feldspathic ceramic, zirconia and lithium disilicate.

The oral hygiene session will be carried out every 6 months (2-years follow-up; 6 sessions), after instruction and motivation of the patient, completion of the clinical chart with the recording of the Probing Depth (evaluation in mm of the peri-implant sulcus taken by a periodontal probe; 4 surfaces of the gingival margin are detected: vestibular, palatal/lingual, mesial, distal), Bleeding on Probing and Plaque Index.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Presence of at least one dental implant
* Good compliance

Exclusion Criteria:

* Patients with cardiac stimulators
* Patients with neurological disorders
* Patients with psychological disorders
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) | Baseline (T0), 6 months (T1), 12 months (T2), 18 months (T3) 24 months (T4)
  Evaluation in mm of the peri-implant sulcus taken by a periodontal probe. 4 surfaces of the gingival margin are detected: vestibular, palatal/lingual, mesial, distal.
Change in Bleeding on Probing (BoP) | Baseline (T0), 6 months (T1), 12 months (T2), 18 months (T3) 24 months (T4)
  Evaluation of the presence or absence of gingival bleeding during a probing with a dichotomous scoring (yes/no) of bleeding sites. The sum of the bleeding sites is divided for the total sites and multiplied per 100.
Change in Plaque Control Record | Baseline (T0), 6 months (T1), 12 months (T2), 18 months (T3) 24 months (T4)
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.